CLINICAL TRIAL: NCT02164799
Title: Establishing a Tool to Increase the Accuracy of Emergency Physicians Diagnosing Etiologies of Shock
Brief Title: The Epidemiology and Approach to Differentiating Etiologies of Shock in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Henning, Instructor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2012P-000357
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Undifferentiated Shock
Keywords: Shock; Predicting diagnosis; Predicting adverse outcomes
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Shock: Patients found to have persistent hypotension after resuscitation or vasopressor requirement
- Pre-shock: Patients with markedly abnormal vital signs (Heart Rate (HR)>130, Respiratory Rate (RR)>24, Shock Index >1, Lactate > 4.0mmol/L, or Systolic Blood Pressure (SBP) <90mm/hg) without shock, as defined previously.

SUMMARY:
The Shock Tool study is designed to improve the clinical evaluation for differentiating shock in the emergency department. The goal of this study is to evaluate and improve the accuracy of physicians differentiating causes of shock.

DETAILED DESCRIPTION:
Specific Aim #1: To study the epidemiology of shock in the emergency department Hypothesis 1: We will better understand shock states if we determine shock etiology among patients presenting to the emergency department in a carefully conducted observational prospective study.

Specific Aim #2: To determine the accuracy of physician diagnosis for the underlying etiology of shock.

Hypothesis 2: Physician assessment of the underlying cause of shock is challenging and often inaccurate in the early stages of care in the emergency department.

Specific Aim #3: To optimize the evidence-based approach to assist in the diagnosis of shock etiology from elements readily available when a patient demonstrates shock physiology in the Emergency Department.

Hypothesis 3: An evidenced-based, standardized approach to clinical decision making integrating elements of the history, physical exam, and early testing will improve a physician's ability to accurately differentiate etiologies of shock.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or great
* For pre-shock cohort: HR > 130, RR>24, Shock index > 1, lactate > 4.0mmol/L, SBP < 90mm/hg)
* For shock cohort: persistent blood pressure <90mm/hg after resuscitation

Exclusion Criteria:

* seizure
* isolated atrial fibrillation with discharge after rate control achieved
* discharged from the emergency department
* intoxication or withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department patients
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Etiology of Shock | Retrospectively, 1 month after enrollment
  Each patient determined to have shock in the emergency department is given a single diagnosis by a reviewing physician after the hospital course is completed.

SECONDARY OUTCOMES:
In hospital mortality | This measure will be assessed at the time of physician review after discharge from hospital, on average 2 months after initial ED visit.
  Death by any cause during hospitalization

OTHER OUTCOMES:
Deterioration | This measure will be assessed at the time of physician review after discharge from hospital, on average 2 months after initial ED visit.
  A composite outcome met if any of the following are present during hospitalization: acute renal failure (creatinine 2x baseline or new initiation of dialysis), non-elective intubation, vasopressor requirement, or mortality.